CLINICAL TRIAL: NCT00002034
Title: A Study of the Safety and Tolerance of Long-Term Therapy With Intravenous Cytovene (Ganciclovir Sodium) for Cytomegalovirus Retinitis in Persons With AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 029F; ICM 1692
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1992-01

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: Retinitis; AIDS-Related Opportunistic Infections; Ganciclovir; Drug Interactions; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome; Zidovudine
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; Retinitis; AIDS-Related Opportunistic Infections; Multiple Acyl Coenzyme A Dehydrogenase Deficiency; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome | interventions — Zidovudine; Ganciclovir

INTERVENTIONS:
Drug: Zidovudine
Drug: Ganciclovir

SUMMARY:
To evaluate the safety and tolerance of long-term ganciclovir (DHPG) therapy for newly diagnosed macular threatening Cytomegalovirus (CMV) retinitis in AIDS patients. To evaluate the clinical response to a 52 week course of intravenous DHPG therapy. To evaluate the safety and tolerance of long-term DHPG with concurrent treatment with zidovudine (AZT). (Patients utilizing treatment with other anti-retroviral drugs will be considered for study entry on a case by case basis.) To determine survival in this group of patients with AIDS and CMV retinitis.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Topical acyclovir.
* Selected cytokines.
* Allowed after the first 4 weeks of ganciclovir:
* Zidovudine (AZT) at a reduced dose (500 mg/day) in patients who have tolerated ganciclovir without grade 3/4 hematological toxicity.
* Other anti-retrovirals after consultation with the Syntex study monitor.

Patients must have the following:

* AIDS and newly diagnosed Cytomegalovirus (CMV) retinitis.
* An understanding of the nature of the study, agreement to its provisions, and willingness to sign the informed consent approved by the appropriate institutions review board, and Syntex.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Have only peripheral CMV retinitis (defined as a lesion outside the major temporal vascular arcades, greater than 1500 microns from the optic disk, or greater than 3000 microns from the fovea).
* Ocular media opacities (corneal, lenticular, or vitreal) preventing ophthalmologic retinal assessment.
* Ocular conditions requiring immediate surgical correction (eg:
* retinal tear or detachment).
* Demonstrated hypersensitivity to acyclovir or ganciclovir.
* Dementia, decreased mentation or other encephalopathic signs and symptoms which would interfere with the ability of the patient to comply with the protocol.

Concurrent Medication:

Excluded:

* Antimetabolites.
* Alkylating agents.
* Nucleoside analogs (excluding selected anti-retroviral agents).
* Imipenem-cilastatin.
* Interferons.
* Selected cytokines.
* Acyclovir (except topical acyclovir).

Patients with the following are excluded:

* Have only peripheral CMV retinitis (defined as a lesion outside the major temporal vascular arcades, greater than 1500 microns from the optic disk or greater than 3000 microns from the fovea).
* Concomitant conditions or diseases described in Exclusion Co-Existing Conditions.

Prior Medication:

Excluded within 1 month of study entry:

* Previous treatment with anti-cytomegalovirus therapy (e.g., ganciclovir, foscarnet or CMV hyperimmune globulin).

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100

CONTACTS AND LOCATIONS:
Locations (9):
- United States (8):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Summitt Med Ctr / San Francisco Gen Hosp, Oakland, California
  - Stanford at Kaiser / Kaiser Permanente Med Ctr, San Francisco, California
  - Miami Veterans Administration Med Ctr, Miami, Florida
  - Dr Winkler Weinberg, Roswell, Georgia
  - SUNY / Health Sciences Ctr at Stony Brook, Stony Brook, New York
  - Dr Alfred F Burnside Jr, Columbia, South Carolina
  - Univ TX Galveston Med Branch, Galveston, Texas
- Southern Alberta HIV Clinic / Foothills Hosp, Calgary, Alberta, Canada